CLINICAL TRIAL: NCT05678322
Title: Optimizing Timing of rhPSMA-7.3 (18F) for Assessing Site(s) of Recurrent Disease Following Radical Prostatectomy
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Blue Earth Diagnostics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22-00547
Record Dates: First submitted 2022-12-28; First posted 2023-01-10 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Patients with PSA > 0.2 ng/ml following Radical Prostatectomy (Experimental): Men will be eligible for the study when their post-prostatectomy PSA level is initially observed to be PSA >0.2ng/ml. All participants will receive a baseline rhPSMA-7.3 (18F) MRI scan within a month of enrollment, and the second rhPSMA-7.3 (18F) scan will be performed within a year of the initial scan. Only those participants with rhPSMA-7.3 (18F) identifiable disease during the initial scan will be offered salvage intervention per standard of care. All participants with a negative initial rhPSMA-7.3 (18F) scan will undergo a second scan when the PSA> 0.5 ng/ml or one year after the initial PET scan. The salvage intervention will be at the discretion of the investigator.
  Interventions: Drug: 18F-Labeled Positron Emission Tomography (PET) Diagnostic Agent; Device: PET MRI Imaging

INTERVENTIONS:
Drug: 18F-Labeled Positron Emission Tomography (PET) Diagnostic Agent — Under development for the diagnosis of prostate cancer by Blue Earth Diagnostics. rhPSMA-7.3 (18F) will be administered intravenously as a single-dose injection. The molecular structure of the drug substance comprises a prostate-specific membrane antigen (PSMA) binding motif, a peptide spacer, an 18F-radiolabeled silicon fluoride acceptor moiety and a gallium chelator complex.
  Other Names: rhPSMA-7.3 (18F)
Device: PET MRI Imaging — rhPSMA-7.3 (18F) PET MRI imaging will be conducted once at baseline and a second time within one year of the initial scan.

SUMMARY:
All men following Radical Prostatectomy (RP) at NYU Langone Health undergo routine prostate specific antigen (PSA) testing in order to identify disease recurrence. By consensus, a BCR following RP occurs once the PSA > 0.2 ng/ml/ Biochemical recurrence often develops years prior to clinical evidence of disease recurrence. Early identification of the site(s) of disease recurrence enables early salvage intervention. Men will be eligible for the study at the point in time their post-prostatectomy PSA level first becomes >0.2 ng/ml. Only those patients with rhPSMA-7.3 (18F) identifiable disease (local, nodal or systemic) will be offered salvage intervention per standard of care. All patients with a negative initial rhPSMA-7.3 (18F) scan will undergo a second scan when the PSA is > 0,5 ng/ml or one year after the initial PET study. The salvage interventions will be at the discretion of the investigator. The study will compare the diagnostic yield of the first and second rhPSMA-7.3 (18F) studies.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients will include all men between age 18 -100 years old,-that have had RP, at the first point in time the PSA > 0.2 ng/ml.

Exclusion Criteria:

* Any contraindication for MRI imaging.
* Prior allergic reaction to rhPSMA-7.3 (18F).
* Patient refuses rhPSMA-7.3 (18F) PET/MRI.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Percentage of Positive PCa Screens | Baseline, Up to Month 24
  This measurement will calculate the change in the percentage of participants who screen positive for prostate cancer (PCa) at the baseline rhPSMA-7.3 (18F) scan vs. the second scan.

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Lepor, MD, Principal Investigator — NYU Langone Medical Center
Locations (1):
- Smilow Comprehensive Prostate Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No